CLINICAL TRIAL: NCT03119571
Title: ACCESS to the Cardiac Catheterization Laboratory in Patients Without ST-segment Elevation Myocardial Infarction Resuscitated From Out-of-hospital Ventricular Fibrillation Cardiac Arrest
Brief Title: ACCESS to the Cardiac Cath Lab in Patients Without STEMI Resuscitated From Out-of-hospital VT/VF Cardiac Arrest
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low enrollment, funding withdrawn
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CV-2017-25768
Record Dates: First submitted 2017-03-29; First posted 2017-04-18 (Actual); Results first posted 2021-01-27 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Cardiac Arrest Due to Underlying Cardiac Condition; Ventricular Fibrillation; Cardiopulmonary Arrest With Successful Resuscitation
Keywords: Cardiac arrest; Ventricular fibrillation; coronary artery disease
MeSH Terms: conditions — Ventricular Fibrillation; Heart Arrest; Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Initial CCL admission (Experimental): Admission to the CCL to evaluate the coronary artery disease
  Interventions: Procedure: Initial CCL admission
- Initial ICU admission (Active Comparator): Admission to the ICU to be evaluated by clinical team and the clinical treatment will be decided by the admitting/attending team.
  Interventions: Diagnostic Test: Initial ICU admission

INTERVENTIONS:
Procedure: Initial CCL admission — Admission to the cardiac catheterization lab to evaluated coronary artery disease and if present fix the culprit lesion/lesions
  Arms: Initial CCL admission
Diagnostic Test: Initial ICU admission — Evaluate for additional testing and/or procedures
  Arms: Initial ICU admission

SUMMARY:
To determine if survival to hospital discharge with good neurological outcome for adults ages 18-75 who are resuscitated from out-of-hospital VT/VF cardiac arrest without clinical signs of a heart attack do better by going straight to the cardiac catheterization laboratory or admitted to the intensive care unit for evaluation. The investigators think a large portion of resuscitated patients presenting with VT/VF have ischemic heart disease which is the cause for the arrest. And prompt access to the cardiac catheterization laboratory to reverse the blocked artery will improve survival with good neurological outcomes.

DETAILED DESCRIPTION:
Primary Aim

Determine survival to hospital discharge with Modified Rankin Scale Score (mRS) ≤ 3 in adult (18-75 years old) patients resuscitated from out-of-hospital VT/VF cardiac arrest who do not have ST-segment elevation on emergency department 12-lead ECG (no-STEMI) randomized to receive either: 1) initial CCL admission, or 2) initial ICU admission.

Hypothesis: The corresponding hypothesis is that a large proportion of all resuscitated patients presenting with VT/VF have ischemic heart disease as the underlying cause for the participants cardiac arrest and that a strategy to facilitate prompt revascularization in all patients presenting with VT/VF who do not have ST-segment elevation on emergency department 12-lead ECG will improve survival with good neurological outcome.

Primary Endpoint

Survival to hospital discharge with mRS ≤ 3

Secondary Aims

Determine secondary assessments of survival, left ventricular function, hospital duration, and rehabilitation in-hospital and assessment of survival and functional status at 3 months in both groups.

Hypothesis: The corresponding hypothesis is that initial CCL admission will result in improved secondary assessment values at 3 months.

Secondary Endpoints

In-hospital secondary endpoints: Survival to hospital discharge, CPC score, mean peak troponin level, mean ejection fraction, mean length of ICU stay, mean hospitalization duration, the incidence of and mean length of rehabilitation.

3-month post-hospital discharge secondary endpoint: Survival to 3 months, survival to 3 months with mRS ≤ 3, functional status at 3 months (CPC score), incidence and length of rehabilitation, incidence of congestive heart failure, incidence of re-hospitalization over 3 months, and incidence and time to return to work.

Pragmatic Clinical Trial

The ACCESS Trial will randomize patients to receive one of two standard treatments currently practiced in the United States: either, 1) initial CCL admission, or 2) initial ICU admission. Other than randomizing to one of these two standard treatments, care is not otherwise specified and is completely at the discretion of the treating clinician, including coronary interventions, if any, hemodynamic support, medications, therapeutic hypothermia, and all other interventions and clinical care.

ELIGIBILITY:
Inclusion Criteria:

* Adult presumed or known to be 18-75 years old
* Resuscitated from OOHCA
* Initial cardiac arrest rhythm of pulseless VT/VF (including patients treated with an AED)
* No ST-segment elevation MI (No STEMI) (or STEMI-equivalent syndrome) on ED 12-lead ECG (as interpreted by a physician)

Exclusion Criteria:

* Initial non-shockable out-of-hospital cardiac arrest rhythm (pulseless electrical activity or asystole)
* Valid do not resuscitate orders (DNR),
* Blunt, penetrating, or burn-related injury, drowning, electrocution or known overdose,
* Known prisoners
* Known pregnancy,
* ST-segment elevation on ED 12-lead ECG (as interpreted by a physician)
* Absolute contraindications to emergent coronary angiography including,
* known anaphylactic reaction to angiographic contrast media,
* active gastrointestinal or internal bleeding, or
* severe concomitant illness that drastically shortens life expectancy or increases risk of the procedure.
* Suspected or confirmed intracranial bleeding
* Refractory cardiac arrest (prior to randomization)
* Patients meeting ACCESS Trial eligibility criteria initially seen in an outside hospital and then transferred to an ACCESS Trial participating hospital

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2017-12-12 (Actual); Primary Completion 2019-11-26 (Actual); Study Completion 2019-11-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Demetris Yannopoulos, MD, Principal Investigator — University of Minnesota; Tom Aufderheide, MD, Principal Investigator — MCW
Locations (23):
- United States (21):
  - Grady Memorial Hospital, Atlanta, Georgia
  - Indiana University Health Methodist Hospital, Indianapolis, Indiana
  - University Hospital, Ann Arbor, Michigan
  - St. Joseph Mercy Hospital, Ypsilanti, Michigan
  - North Memorial Medical Center, Brooklyn Center, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - University of Minnesota Medical Center, Fairview, Minneapolis, Minnesota
  - Methodist Hospital, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - St. Joseph's Hospital, Saint Paul, Minnesota
  - University of Cincinnati, Cincinnati, Ohio
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Miriam Hospital, Providence, Rhode Island
  - Rhode Island Hospital, Providence, Rhode Island
  - Parkland Memorial Hospital, Dallas, Texas
  - University of Utah, Salt Lake City, Utah
  - Virginia Commonwealth University Hospital, Richmond, Virginia
  - Harborview Medical Center, Seattle, Washington
  - Medical College of Wisconsin Froedtert Hospital, Milwaukee, Wisconsin
- Canada (2):
  - St. Paul's Hospital, Vancouver, British Columbia
  - Vancouver General Hospital, Vancouver, British Columbia

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Initial CCL Admission | Initial ICU Admission
Started | 31 | 34
Completed | 31 | 34
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Initial CCL Admission | Initial ICU Admission | Total
Number analyzed (Participants) | 31 | 34 | 65
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 22 | 22 | 44
  >=65 years | 9 | 12 | 21
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 13 | 21
  Male | 23 | 21 | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 24 | 24 | 48
  Unknown or Not Reported | 6 | 9 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 6 | 4 | 10
  Black or African American | 0 | 0 | 0
  White | 20 | 29 | 49
  More than one race | 4 | 1 | 5
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Canada | 0 | 1 | 1
  United States | 31 | 33 | 64

OUTCOME MEASURES:

1. Primary Outcome: Survival to Hospital Discharge With mRS ≤ 3
Description: Outcome is reported as the percent of participants who survive to hospital discharge with an mRS score less than or equal to 3. The Modified Rankin Score (mRS) is a 6-point scale measuring disability. Scores range from 0 (no disability) to 5 (severe disability; bedridden, incontinent, requires continuous care). Higher scores indicate greater disability. A sixth category is often added for patients who expire.
Time Frame: Up to 3 weeks
Population: Of the 34 participants in the ICU group, 27 survived to discharge and 7 died. Of the 31 participants in the CCL group, 24 survived to discharge, and 7 died.
Measure: Number; unit: percentage of participants
Arm/Group | Initial CCL Admission | Initial ICU Admission
Number analyzed (Participants) | 24 | 27
percentage of participants | 67.7 | 73.5

ADVERSE EVENTS:
Time Frame: Length of hospitalization, up to 3 weeks
Description: Before the trial started, a list of predefined adverse events was written in the study protocol for both groups. These events fall into 7 categories that were expected for this population. No additional adverse events were collected.
Arm/Group | Initial CCL Admission | Initial ICU Admission
All-Cause Mortality (participants affected / at risk) | 7/31 | 7/34
Serious Adverse Events (participants affected / at risk) | 12/31 | 18/34
Other Adverse Events (participants affected / at risk) | 0/31 | 0/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Initial CCL Admission (N=31) | Initial ICU Admission (N=34)
Infection/sepsis (Infections and infestations) | 9 (15) | 11 (16)
Acute Kidney Injury (Renal and urinary disorders) | 4 (4) | 7 (7)
Liver Failure/Injury (Hepatobiliary disorders) | 1 (1) | 2 (2)
Cardiogenic Shock (Cardiac disorders) | 7 (10) | 5 (5)
Multiple Organ Dysfunction Syndrome (MODS) (General disorders) | 1 (2) | 1 (2)
Seizure Activity (Nervous system disorders) | 2 (2) | 3 (3)
Cardiac Arrest (Cardiac disorders) | 4 (4) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2018-10-25): https://cdn.clinicaltrials.gov/large-docs/71/NCT03119571/Prot_SAP_000.pdf
  • Informed Consent Form: Main Consent (2019-01-03): https://cdn.clinicaltrials.gov/large-docs/71/NCT03119571/ICF_001.pdf
  • Informed Consent Form: Continued Participation Consent (2019-01-03): https://cdn.clinicaltrials.gov/large-docs/71/NCT03119571/ICF_002.pdf